CLINICAL TRIAL: NCT03804385
Title: Primary Spontaneous Pneumothorax and Different Types of Surgical Management
Brief Title: Surgical Management of Primary Spontaneous Pneumothorax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed samir yussef, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pneumothoracic
Record Dates: First submitted 2018-05-09; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intercostal tube (Other): insertion of intercostal tube is surgical operation used in pneumothorax
  Interventions: Procedure: intercostal tube

INTERVENTIONS:
Procedure: intercostal tube — surgical operation

SUMMARY:
the different surgical management in patients with primary pneumothorax 0 Objective 1: Identify risk factors that are predictive of the need for surgical intervention.

* Objective 2: Determine the value of management strategies in terms of hospital stay
* Objective 3: Assess outcomes and postoperative results including symptom relive ,or recurrence or post-operative complications .

DETAILED DESCRIPTION:
pneumothorax is defined as air or gas accumulated in the pleural cavity. Spontaneous pneumothorax can be classified as either primary or secondary. Primary spontaneous pneumothorax , which is defined as a pneumothorax without underlying lung disease, predominantly occurs in young, thin males. It is usually caused by ruptured pleural blebs or bullae. Secondary spontaneous pneumothorax usually occurs in older people with underlying pulmonary disease, such as emphysema or asthma, acute or chronic infections, lung cancer, and congenital diseases including cystic fibrosis, catamenial pneumothorax , or lymphangio-leiomyomatosis .

The age-adjusted incidence of Primary spontaneous pneumothorax is from 7.4 to 18 per 100 000 population per year in males, and from 1.2 to 6 per 100 000 population per year in females. It usually occurs in tall, thin males of 10 to 30 years old. Less often does it occur in people at the age of more than 40 years. Primary spontaneous pneumothorax might be associated with some congenital disorders such as Marfan's syndrome, or some environmental factors such as smoking. Primary spontaneous pneumothorax usually occurs at rest. Approximately 10% of patients with Primary spontaneous pneumothorax have a positive family history. Smoking is also regarded as a precipitating factor for Primary spontaneous pneumothorax. The relative risk of pneumothorax ranged from 7 to 100 times higher in light to heavy smokers Most authors believe that Primary spontaneous pneumothorax results from spontaneous rupture of a sub-pleural bleb or bulla. However, only a portion of patients with Primary spontaneous pneumothorax could be found with blebs or bullae in imaging or at the time of surgery. Other mechanisms may be considered, such as increase in pleural porosity secondary to inflammation. The development of bullae, blebs, or pleural porosity might be related to many factors, such as distal airway inflammation, distal bronchial tree anomaly, disorders of connective tissue formation, local ischemia, and malnutrition.

Primary spontaneous pneumothorax usually occurs at rest, and presents with acute onset of local pleuritic chest pain accompanied by dyspnoea. This pain may be mild or severe, sharp and steady ache in character, and usually resolves within 24 h even though pneumothorax still exists. On physical examination, decreased air entry on auscultation, decreased chest wall movement on inspection, hyper-resonance (tympanic) on percussion are most often detected in patients with large pneumothorax (free air occupies more than 15% to 20% area of hemi thorax). Reflex tachycardia can be found in most patients in response to discomfort or circulating or respiratory compromise. Tension pneumothorax should be suspected if severe tachycardia, cold sweating, hypotension, or cyanosis has developed. Blood gas analysis in patients with large pneumothoraces may reveal increased alveolar-arterial difference in oxygen partial pressure (PA-aO2) due to increased intrapulmonary shunt from the collapsed lung.

Most Primary spontaneous pneumothorax cases are confirmed by upright posteroanterior chest radiograph, which can be used to assess the pneumothorax size with good accuracy. A pleural line with or without an air-fluid level can be seen in the chest radiograph, but sometimes it is difficult to detect these signs, especially in patients with small pneumothoraces, emphysema, or poor exposure of the film. Expiratory chest radiographs have no diagnostic value for patients with Primary spontaneous pneumothorax.

Computed tomography (CT) of the chest can be used to detect patients with small penman-thorax (less than 15% area of hemi thorax). In addition, CT can provide more detailed information to assist in the subsequent management. Findings which can be noted include the number, size, and location of bullae/blebs (ipsi- or contra-laterally), as well the possibilities of pleural adhesion, pleural fluid accumulation, and possible underlying pulmonary diseases. For more than 90% of patients with Primary spontaneous pneumothorax, pathological lung changes can be detected by CT. The most common type is few (n<5) and small (<2 cm in diameter) blebs, followed by mixed blebs and bullae (>2 cm in diameter).

The first line of management of primary spontaneous pneumothorax is intercostal tube insertion .that provide management of this case and only recurrent or persisting cases need further surgical management.

Surgical management of Primary spontaneous pneumothorax is usually indicated in patients with recurrent ipsi-lateral pneumothorax, first episode with occupational risk or persistent air-leakage (more than 5 to 7 d), or prior contra-lateral pneumothorax. A first episode of a Primary spontaneous pneumothorax is treated by observation if the area of pneumothorax is <20% or by simple aspiration if >20%, but recurrences are frequent. For recurrent or persisting pneumothorax, a more invasive surgical approach is indicated. The procedure can be approached through open thoracotomy or video-assisted thoracic surgery.

There are two objectives in the surgical management of pneumothorax. The first widely accepted objective is resection of blebs or the suture of apical perforations to treat the underlying defect. The second objective is to create a pleural symphysis to prevent recurrence. There is nearly zero mortality and very low major morbidity with either video-assisted thoracic surgery or open approaches. Postoperative complications are low (5%-10%), and usually minor and self-limited, including prolonged air-leakage, pleural effusion or hemorrhage, wound infection or hematoma, pulmonary atelectasis or pneumonia.

The traditional open approach has gradually been replaced by minimally invasive video-assisted thoracic surgery in the diagnosis and treatment for patients with various intrathoracic diseases, including the treatment of Primary spontaneous pneumothorax. The outcomes of video-assisted thoracic surgery for patients with Primary spontaneous pneumothorax are very good compared to conservative treatment and equal to those of open thoracotomy. The video-assisted thoracic surgery approach has the benefits of less postoperative pain, better wound cosmetics, shorter hospital stay and duration of drainage, better functional recovery, better short and long term patient satisfaction, and equivalent cost-effectiveness to the open approach.video-assisted thoracic surgery is recommended as the first-line surgical treatment for patients with recurrent Primary spontaneous pneumothorax or first episode of Primary spontaneous pneumothorax. However, the recommendation can only be graded as B or C as there have been only a limited number of patients in relevant randomized trials.

The risk of postoperative recurrence requiring re-operation for the video-assisted thoracic surgery and surgical groups varies in different reported series. However, re-operation following video-assisted thoracic surgery is more often required than that after open thoracotomy, with a higher rate of both late recurrent pneumo-thorax and prolonged early postoperative air-leakage.

video-assisted thoracic surgery for Primary spontaneous pneumothorax can be accomplished mostly through three ports, but two or single port(s) with the use of single incision port laparoscopic surgery (SILS) system has been reported in recent years. Endotracheal general anesthesia with the use of a double or single lumen endotracheal tube is still recommended by most reported series for Primary spontaneous pneumothorax patients undergoing video-assisted thoracic surgery . video-assisted thoracic surgery procedures through local or epidural anesthesia for patients with Primary spontaneous pneumothorax (the awake procedure) have been reported The bullae/blebs in patients with Primary spontaneous pneumothorax can be managed through video-assisted thoracic surgery by stapling and resection, no-knife stapling, suturing, or endo-loop ligation. Pleurodesis is usually required in addition to bullae/blebectomy for surgical management of patients with Primary spontaneous pneumothorax. It can significantly decrease the risk of early air-leakage or late recurrence, which is especially important for patients undergoing video-assisted thoracic surgery .

Since the surgical treatment for patients with Primary spontaneous pneumothorax has become less invasive through video-assisted thoracic surgery in recent years, there have been many published papers suggesting the use of this surgical intervention for patients with the first Primary spontaneous pneumothorax There are still some reported series that do not agree with the use of video-assisted thoracic surgery after the first Primary spontaneous pneumothorax. Retrospective cost effective analysis has revealed that tube thoracostomy should be used at first occurrence, followed by video-assisted thoracic surgical bullae/blebectomy and pleurodesis in case of recurrence. However, these studies were only based on single, retrospective, and small case number analyses, and the patient satisfaction and quality of life were not considered. video-assisted thoracic surgery will be expected as an option of management for patients with their first Primary spontaneous pneumothorax. However, the management of the first Primary spontaneous pneumothorax remains controversial because there is still little high-quality evidence to guide the decision-making

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with primary pneumothorax at Assiut University Hospital patients above 18 years and less 40 years Male or Females

Exclusion Criteria:

Patients with other chest pathology including :

* emphysema
* asthma,
* acute or chronic infections
* lung cancer,
* congenital diseases including( cystic fibrosis, catamenial pneumothorax, or lymphangioleiomyomatosis)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Duration of Intercostal tube in days | 2 weeks
  last more in open thoracotomy
Duration of air leakage in days | 2 weeks
  last more in intercostal tube than in open thoracotomy
recurrence after one year | one year
  by radiological intervention on after one year follow up
pain score | 1 week
  high pain score in open thoracotomy than in intercostal tube

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine Assiut Univeresity, Asyut
  - School of Medicine Assiut Univeresity, Asyut